CLINICAL TRIAL: NCT00982033
Title: A Randomized, Blinded, Placebo-Controlled Six Month Treatment Trial of Aliskiren to Improve Exercise Tolerance in Older Patients With Heart Failure and Normal Ejection Fraction
Brief Title: Effects of Aliskiren on Patient With Heart Failure and a Normal Ejection Fraction
Acronym: Aliskiren
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00008625; CTA study # CSPP100AUS13T; GTS # 34136
Record Dates: First submitted 2009-09-18; First posted 2009-09-22 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Heart failure with normal ejection fraction; Elderly
MeSH Terms: conditions — Heart Failure | interventions — aliskiren

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Aliskiren (Active Comparator): 50 % of subjects participating in this trial will be on the active medication, Aliskiren 300mg qd, the other 50% will be on placebo.
  Interventions: Drug: aliskiren
- Placebo (Placebo Comparator): 50% of subjects will be randomized to placebo.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: aliskiren — aliskiren 300mg qd versus placebo for 24 weeks.
  Other Names: Tekturna
  Arms: Aliskiren
Drug: placebo — placebo qd for 24 weeks
  Arms: Placebo

SUMMARY:
The primary objective of this study is to determine whether treatment with aliskiren (300 mg) compared to placebo will improve treadmill exercise time in older (age ≥ 55 years) patients with heart failure and normal ejection fraction (HFNEF).

DETAILED DESCRIPTION:
Heart Failure with Normal Ejection Fraction (HFNEF) is the most common form of heart failure, particularly in older persons. However, the optimal therapy for this disorder has not been defined. The primary chronic symptom in HFNEF is exercise intolerance, manifested by shortness of breath and fatigue with exercise. This is the major determinant of quality of life, can be measured objectively and reproducibly and is modifiable.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 55 years of age
* Symptomatic HFNEF of at least 1 month duration.
* Reduced early diastolic mitral annular velocity by tissue Doppler
* Left ventricular ejection fraction (LVEF ≥ 0.50)
* Baseline exercise intolerance
* Patients who are able to provide written informed consent
* Stable medical therapy for 30 days prior to screening

Exclusion Criteria:

* Seated blood pressure ≥ 160/90 mmHg at Visit 1 (screening)
* Clinically significant pulmonary disease
* Known history of documented EF < 0.45 at any time
* Clinically unstable heart failure, medication changes for worsening heart failure symptoms within the past 4 weeks
* Severe anemia (Hgb <10 mg/dL)
* Clinical evidence of uncontrolled hypo or hyperthyroidism
* Clinically significant valvular heart disease
* Surgical correction of valvular heart disease within the last year
* Known familial hypertrophic cardiomyopathy or hypertrophic obstructive cardiomyopathy
* Known restrictive cardiomyopathy or systemic illness known to be associated with infiltrative myocardial disease (e.g. amyloidosis, sarcoidosis, hemachromatosis)
* Pericardial restriction or hemodynamically significant pericardial effusion
* Cor pulmonal or other causes of right heart failure not related to LV dysfunction
* Extreme obesity (weight > 325 pounds)
* Acute coronary syndrome within past 3 months
* Coronary artery revascularization within past 3 months
* Peripheral artery revascularization within past 3 months
* Acute cerebrovascular syndrome (stroke or TIA) within the past 3 months
* Uncontrolled symptomatic brady- or tachyarrhythmia
* Creatinine > 2.5 mg/dl at screening
* Potassium > 5.2 meq/l at screening
* Prior treatment with, hypersensitivity to, intolerance of or contra-indication to aliskiren
* Current treatment with antidepressant medication in the MAO(Monoamine Oxidase) inhibitor or SSRI(Selective serotonin reuptake inhibitors) class
* Current participation in another clinical trial
* Current treatment with both an ACE(Angiotensin-converting enzyme) inhibitor and an angiotensin receptor antagonist.
* Known significant bilateral renal artery stenosis
* Serious non-cardiovascular disease severely limiting life expectancy
* Previous major organ (e.g., lung, liver, heart, kidney) transplantation or on a transplant waiting list
* Any condition that is likely to prevent the patient from complying with the requirements of the study or completing the study (e.g., history of poor compliance, alcohol or drug dependency, psychiatric illness, no permanent home)
* Pregnant women, nursing women, and women of childbearing potential.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-07; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Scott JM, Haykowsky MJ, Eggebeen J, Morgan TM, Brubaker PH, Kitzman DW. Reliability of peak exercise testing in patients with heart failure with preserved ejection fraction. Am J Cardiol. 2012 Dec 15;110(12):1809-13. doi: 10.1016/j.amjcard.2012.08.015. Epub 2012 Sep 13. PMID 22981266
- [Derived] Upadhya B, Brubaker PH, Morgan TM, Eggebeen JD, Jao GT, Stewart KP, Kitzman DW. The effect of Aliskiren on exercise capacity in older patients with heart failure and preserved ejection fraction: A randomized, placebo-controlled, double-blind trial. Am Heart J. 2018 Jul;201:164-167. doi: 10.1016/j.ahj.2018.03.019. Epub 2018 Apr 4. PMID 29910050

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren | Placebo
Started | 25 | 27
Completed | 25 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Aliskiren: 50 % of subjects participating in this trial will be on the active medication, Aliskiren 300mg qd.
  aliskiren: aliskiren 300mg qd for 24 weeks.
- Placebo: 50% of subjects participating in this trial will be randomized to placebo.
  placebo: placebo qd for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Aliskiren | Placebo | Total
Number analyzed (Participants) | 25 | 27 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (6.3) | 70.6 (7.7) | 69.9 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Exercise Treadmill Time
Description: Treadmill exercise time to exhaustion on the modified naughton protocol.
  LS-mean is in effect, within-group means appropriately adjusted for the other effects in the model.
Time Frame: Baseline, 24 week visit
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Aliskiren | Placebo
Number analyzed (Participants) | 25 | 27
seconds
  Baseline | 621 (120) | 580 (126)
  24 Week | 624 (151) | 579 (145)
  LS Mean | 607 (13) | 605 (12)
Statistical Analysis 1: Comparison: Aliskiren vs Placebo; Test type: Superiority or Other; p = 0.90, ANCOVA

ADVERSE EVENTS:
Time Frame: 2 years, 2 months
Arm/Group | Aliskiren | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 4/27
Other Adverse Events (participants affected / at risk) | 6/25 | 13/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=25) | Placebo (N=27)
dyspnea, CHF exacerbation (Cardiac disorders) | 0 (0) | 2 (2) — Hospitalized for dyspnea, CHF exacerbation
small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) — Surgery for small bowel obstruction.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aliskiren (N=25) | Placebo (N=27)
leg, back and or joint pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
altered mental status (Nervous system disorders) | 0 (0) | 2 (2)
root canal (Surgical and medical procedures) | 0 (0) | 1 (1)
increased blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
pneumonia and or upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
abdominal pain, colitis, and or virus (Gastrointestinal disorders) | 1 (1) | 2 (2)
ear and or eye infection (Ear and labyrinth disorders) | 1 (1) | 1 (1)
viral symdrom and or possible thrush (Endocrine disorders) | 1 (1) | 0 (0)
atrial fibrillation and or palpitations (Cardiac disorders) | 1 (1) | 1 (1)
numbness in left arm (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days